CLINICAL TRIAL: NCT01630590
Title: An Observational Study of XL-184 Cabozantinib and Androgen Ablation in Patients With Androgen-Dependent Metastatic Prostate Cancer
Brief Title: Cabozantinib and Androgen Ablation in Patients With Androgen-Dependent Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Exelixis (Industry); High Impact Clinical Research Support Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0252; NCI-2014-00934 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Results first posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Metastatic Prostate Cancer; Prostate adenocarcinoma; Androgen-Dependent Prostate Cancer; Cabozantinib; XL 184; Androgen Ablation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cabozantinib + Androgen Ablation Therapy (Experimental): Patients receive Cabozantinib at starting dose of 60 mg by mouth every day. Study cycles 3 weeks in duration. Patients stay on treatment as long as they are benefitting. Patients receive androgen ablation therapy, either by means of luteinizing hormone-releasing hormone super-agonist (of any formulation), LHRH antagonist, or surgical castration. Study doctor will decide what hormone therapy patient will receive.
  Interventions: Drug: Cabozantinib; Drug: Androgen Ablation Therapy

INTERVENTIONS:
Drug: Cabozantinib — Starting dose of 60 mg by mouth every day of a 21 day cycle.
  Other Names: XL 184
Drug: Androgen Ablation Therapy — Androgen ablation therapy, either by means of luteinizing hormone-releasing hormone super-agonist (of any formulation), LHRH antagonist, or surgical castration given upon decision of study doctor.

SUMMARY:
The goal of this clinical research study is learn if adding cabozantinib (also known as XL184) to hormonal therapy can help to control prostate cancer. The safety of this drug will also be studied.

Cabozantinib is designed to block certain proteins in your blood that cause cancer cells to grow. This may cause cancer cells to die.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will take 1 capsule of cabozantinib by mouth 1 time every day while you are on study. You should not eat or drink anything other than water for 2 hours before and 1 hour after taking the study drug. You should take the capsule with at least 1 cup (8 ounces) of water. You will also be given separate directions about how to take the study drug.

You will also receive hormone therapy. The hormone drug you receive will be standard of care hormone therapy. The study doctor will decide what hormone therapy you will receive and will explain when and how you should take the hormone therapy, as well as its risks.

You will be given a drug diary where you will record when you take cabozantinib. You should return this diary to the study staff when you come into the clinic.

Study Visits:

At every visit, you will be asked about any side effects you may have had and any other drugs you may be taking.

If you are receiving Coumadin, every week for the first 3 weeks, you will have blood drawn (about 1 teaspoon) to test your blood clotting function.

Every 3 weeks for the first 12 weeks of the study, and then every 6 weeks after that:

* You will have a physical exam.
* Blood (about 3-4 teaspoons) will be drawn for routine tests.

Every 3 weeks for the first 12 weeks of the study, and then every 12 weeks after that, blood (about 1 teaspoon) will be drawn to check your thyroid and pancreatic function. The frequency of the testing may change if the study doctor thinks it is needed.

Every 6 weeks, you will have the following tests performed:

* Blood (about 2-3 teaspoons) will be drawn to measure your PSA levels and for biomarker testing.
* Urine will be collected for routine tests.
* You may have these test performed near your home if the study doctor thinks you are tolerating the treatment.

Every 12 weeks, you will have a bone scan and CT scans of the chest, abdomen, and pelvis to check the status of the disease.

Length of Study:

You may continue receiving the study drug for as long as the study doctor thinks it is in your best interest. You will be taken off study early if the disease gets worse, if you have intolerable side effects, or if your study doctor thinks it is in your best interest to stop.

Long-Term Follow-Up:

You will be contacted every 6 months after you stop taking the study drug to check on how you are feeling and the status of the disease. This will consist of a phone call, e-mail, or medical record review. If you are called, each call should last about 5 minutes.

This is an investigational study. Cabozantinib is FDA approved to treat patients with certain types of thyroid cancer. Its use in this study is investigational.

Up to 60 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic proof of prostate adenocarcinoma
2. Newly diagnosed Androgen-Dependent Prostate Cancer. Patients already on ADT are eligible as long as the time from initiation of LHRH analog or antagonist is not greater than 3 months.
3. Metastatic disease on bone scan and/or involvement of soft tissues (lymph nodes and/or viscera) by CT scan, PET/CT, or MRI
4. PSA > 1 ng/ml, unless anaplastic features are present (according to eligibility 10)
5. Life expectancy from a co-morbid illness > 3 years
6. Eastern Cooperative Oncology Group (ECOG) performance status </= 2
7. Patients must have adequate organ function as defined by: Absolute Neutrophil Count (ANC) >/= 1,500/ul (unless due to bone marrow infiltration by tumor in which case ANC >/=500/ml are allowed) Hemoglobin (Hgb) >/= 9 gm/dL (unless due to bone marrow infiltration by tumor in which case Hgb>8 gm/dL); Total bilirubin </= 1.5times the upper limit of normal (ULN). For patients with known Gilbert's disease, total bilirubin should be </= 3mg/dL; platelet count >/= 100,000/mm^3 (unless due to bone marrow infiltration by tumor in which case >/=50,000/ml are allowed); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) </= 3.0 x ULN if no liver involvement, or </= 5 x ULN with liver involvement; Lipase < 2 x the upper limit of normal; Urine protein/creatinine ratio (UPCR) </= 1; Serum phosphorus >/= lower limits of normal (LLN); estimated creatinine clearance of >/=40 ml/min.
8. Prior ADT is allowed if it was an adjunct to definite local therapy, was given for </=1 year and was completed at least 12 months before initiating therapy for metastatic disease.
9. Prior therapy with other tyrosine kinase inhibitors (TKI) inhibitors or any other type of investigational agent is allowed if it was an adjunct to definitive local therapy, was given for </=6 months, and was completed at least 12 months before initiating therapy for metastatic disease.
10. Patients with "anaplastic" features are eligible for this trial as defined by at least one of the following: a) Any of the following metastatic presentations: exclusive visceral metastases, radiographically predominant lytic bone metastases identified by plain X-ray or CT scan, bulky (>5 cm in longest dimension) lymphadenopathy or high-grade (gleason >8) tumor mass in the prostate/pelvis.; b) Low PSA (</= 10 ng/ml) at initial presentation (prior to androgen ablation or at symptomatic progression in the castrate-setting) plus high volume (>/=20) bone metastases.; c) Elevated serum LDH (>/= 2 x ULN) or elevated serum CEA (>/= 2 x ULN) in the absence of other etiologies.; d) Short interval (</= 180 days) to castrate-resistant progression following initiation of hormonal therapy.
11. Sexually active fertile subjects, and their partners, must agree to use medically accepted methods of contraception (eg, barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of study drug(s).

Exclusion Criteria:

1. Biological agents (antibodies, immune modulators, cytokines, or vaccines) or radionuclide treatment within 6 weeks of the first dose of study treatment.
2. Radiation therapy within 2 weeks prior to initiation of study treatment.
3. Symptomatic or uncontrolled brain metastasis or epidural disease requiring current treatment including steroids and anti-convulsant.
4. The subject has had another diagnosis of malignancy requiring systemic treatment within the last two years, unless non-melanoma skin cancer, or superficial bladder cancer.
5. The subject has uncontrolled or significant intercurrent illness including, but not limited to, the following conditions: Chronically uncontrolled hypertension, defined conventionally as consistent and repeated systolic pressures above 140 mmHg or diastolic pressures above 90 mmHg despite anti-hypertensive therapy. This may be better established with home BP readings than with clinic visit results. There is no criterion related to a specific BP result required for eligibility, nor are acute BP elevations that are related to iatrogenic causes, acute pain, or other transient reversible causes considered to be an exclusion criteria. The intent is to exclude patients with chronically uncontrolled hypertension that might be further exacerbated by Cabozantinib.
6. Continued from # 5) Other cardiovascular disorders such as symptomatic congestive heart failure (CHF), unstable angina pectoris, clinically-significant cardiac arrhythmias, history of stroke (including transient ischemic attack [TIA], or other ischemic event) within 6 months of study treatment, myocardial infarction within 6 months of study treatment, history of thromboembolic event requiring therapeutic anticoagulation within 6 months of study treatment or main portal vein or vena cava thrombosis or occlusion. ;Gastrointestinal (GI) disorders particularly those associated with a high risk of perforation or fistula formation including: Any of the following at the time of screening; a) intra-abdominal tumor/metastases invading GI mucosa b) active peptic ulcer disease, c) inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
7. Continued from # 6) Any of the following within 6 months before the first dose of study treatment: a) history of abdominal fistula b) gastrointestinal perforation c) bowel obstruction or gastric outlet obstruction; d) intra-abdominal abscess. Note: Complete resolution of an intra-abdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more that 6 months ago. GI surgery (particularly when associated with delayed or incomplete healing) within 28 days. Note: Complete healing following abdominal surgery must be confirmed prior to initiating treatment with cabozantinib even if surgery occurred more that 28 days ago. Other disorders associated with a high risk of fistula formation including PEG tube placement within 3 months before the first dose of study therapy or concurrent evidence of intraluminal tumor involving the trachea and esophagus.
8. The subject is unable to swallow capsules tablets
9. The subject has a previously-identified allergy or hypersensitivity to components of the study treatment formulation.
10. Oral corticosteroids >/= 7.5mg/day prednisone (or prednisone equivalents).
11. Prior treatment with cabozantinib.
12. The subject has a corrected QT interval calculated by the Fridericia formula (QTcF) >500 ms within 28 days before randomization.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-01-08 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Corn, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from January 2014 - January 2016 at MD Anderson Cancer Center
Period: Overall Study
Arm/Group | Cabozantinib + Androgen Ablation Therapy
Started | 62
Completed | 5
Not Completed | 57
Not completed — Adverse Event | 9
Not completed — Lack of Efficacy | 37
Not completed — Withdrawal by Subject | 4
Not completed — 2nd primary tumor | 2
Not completed — Automobile accident | 1
Not completed — Maximum benefit | 4

BASELINE CHARACTERISTICS:
Arm/Group | Cabozantinib + Androgen Ablation Therapy
Number analyzed (Participants) | 62
Age, Continuous [Median (Full Range); unit: years] | 62 [47 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 56
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 57
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 62
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG measure a participant's daily living abilities. All participants in this trial are grade 0, grade 1, or grade 2.
  Grade 0: Fully active on all pre-disease performance without restriction Grade 1: light housework and office work. Restricted in physically strenuous activity Grade 2: Ambulatory and capable of self-care. Not able to carry out work that is light or sedentary.
  Participants
    Grade 0 | 45
    Grade 1 | 17
    Grade 2 | 0
Prior Treatment of Primary Tumor [Count of Participants; unit: Participants]
  No Prior Treatment | 46
  Yes Prior Treatment | 16
Gleason Score [Count of Participants; unit: Participants] — Gleason score grades prostate cancer based on the severity of the cancer The scores range from 2 -10. The higher the score the more severe the cancer. Gleason Score of 6 is the lowest cancer grade. In this trial, participants who have a traditional Gleason 7 score with an additional area in the prostate that meets Gleason 5 score were counted separately and labeled Gleason 7 + 5.
  Participants
    Gleason 6-7 | 10
    Gleason 7 + 5 | 2
    Gleason 8-10 | 45
    Unknown Gleason Score | 5
Prostate Specific Antigen (PSA) Levels [Median (Full Range); unit: ng/mL] — PSA is produced by normal and cancerous prostate tissue. PSA levels are often elevated in men with prostate cancer.
  ng/mL | 64.7 [1.2 to 131.6]
Bone Specific Alkaline Phosphatase Level [Median (Full Range); unit: µg/L] — Population: Only 59 of the participants had bone specific Alkaline Phosphatase level as baseline
  µg/L
    number analyzed (Participants) | 59
    (all) | 61 [8.4 to 2000]
Bone Metastases [Count of Participants; unit: Participants] — Bone metastases measures help define the extent on the prostate cancer in the participants. The first measure, Bone Metastases counted the number of participants with bone metastasis. The second measure, Bone Only, counted the number of patients who only had prostate cancer present in the bone.
  Participants
    Bone Metastases | 58
    Bone Only | 27
Visceral Metastases [Count of Participants; unit: Participants] — Visceral Metastases measurement determined how many participants at baseline had prostate tumors in any of the organs of the body. This measurement did not include bone or lymph nodes.
  Participants | 8
Soft-Tissue Metastases [Count of Participants; unit: Participants]
  None | 29
  Lymph Nodes | 33
  Liver | 2
  Lung | 6
Volume of Metastases [Count of Participants; unit: Participants] — The volume of metastases was categorized as high or low. A high volume was defined as a participant who had 3 or more bone tumors and/or visceral tumors.
  Participants
    Low | 8
    High | 54

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression defined by any of the following: (a) radiographic progression (using RECIST 1.1 for visceral disease and PCWG2 for Bone Scans), (b) receive additional anti-cancer therapy, or (c) clinical progression resulting in stopping the treatment.
Time Frame: 31.2 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib + Androgen Ablation Therapy
Number analyzed (Participants) | 62
months | 16.1 [14.6 to 22.7]

2. Primary Outcome: Serious Adverse Events and Other (Not Including Serious) Adverse Events
Description: Number of instances of Serious Adverse Events and Other (Not Including Serious) Adverse Events. Adverse events were monitored for 30 days beyond the last day of treatment. These adverse events are documented. The adverse events are reported as Serious Adverse Events and Adverse Events. Serious Adverse Events are defined as adverse events in which the participant dies, is hospitalized, is disabled, or is exposed to the medicine while pregnant resulting in and birth defect. Adverse events evaluated for all treated participants using the NCI CTCAE version 4.3.
Time Frame: Start of treatment up to 30 days after study drug, up to 80 months
Measure: Number; unit: adverse events
Arm/Group | Cabozantinib + Androgen Ablation Therapy
Number analyzed (Participants) | 62
adverse events
  Other (Not Including Serious) Adverse Events | 2105
  Serious Adverse Events | 3

ADVERSE EVENTS:
Time Frame: From the first dose through 30 days after the last day of treatment, up to 80 months
Arm/Group | Cabozantinib + Androgen Ablation Therapy
All-Cause Mortality (participants affected / at risk) | 24/62
Serious Adverse Events (participants affected / at risk) | 3/62
Other Adverse Events (participants affected / at risk) | 62/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib + Androgen Ablation Therapy (N=62)
Diarrhea (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib + Androgen Ablation Therapy (N=62)
Abdominal Pain (Gastrointestinal disorders) | 6 (8)
Alanine Aminotransferase Increase (Investigations) | 50 (116)
Alkaline Phosphatase Increase (Investigations) | 17 (30)
Alopecia (Skin and subcutaneous tissue disorders) | 15 (17)
Anemia (Blood and lymphatic system disorders) | 41 (56)
Anorexia (Metabolism and nutrition disorders) | 18 (26)
Aspartate Aminotransferase Increase (Investigations) | 52 (148)
Bloating (Gastrointestinal disorders) | 3 (4)
Bilirubin Increase (Investigations) | 11 (16)
Constipation (Gastrointestinal disorders) | 22 (36)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 46 (142)
Dizziness (Nervous system disorders) | 10 (11)
Dry Mouth (Gastrointestinal disorders) | 8 (8)
Dry Skin (Skin and subcutaneous tissue disorders) | 20 (21)
Dysgeusia (Nervous system disorders) | 37 (49)
Dyspepsia (Gastrointestinal disorders) | 7 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19 (26)
Edema (General disorders) | 54 (120)
Fatigue (General disorders) | 54 (120)
Flatulence (Gastrointestinal disorders) | 5 (5)
Flushing (Vascular disorders) | 3 (3)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 18 (25)
Headache (Nervous system disorders) | 7 (8)
Hematuria (Renal and urinary disorders) | 4 (4)
Lactate Dehydrogenase Increase (Hepatobiliary disorders) | 31 (58)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 21 (25)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (16)
Hypernatremia (Metabolism and nutrition disorders) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 8 (8)
Hypertension (Vascular disorders) | 25 (37)
Hyperthyroidism (Endocrine disorders) | 6 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 18 (36)
Hypocalcemia (Metabolism and nutrition disorders) | 8 (12)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 8 (10)
Hypomagnesemia (Metabolism and nutrition disorders) | 31 (67)
Hyponatremia (Metabolism and nutrition disorders) | 5 (8)
Hypothyroidism (Endocrine disorders) | 41 (57)
Lipase Increase (Investigations) | 15 (21)
Memory Impairment (Nervous system disorders) | 3 (3)
Mucositis Oral (Gastrointestinal disorders) | 18 (37)
Cramping in Extremities (Musculoskeletal and connective tissue disorders) | 7 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 21 (57)
Neutrophil Count Decrease (Investigations) | 21 (45)
Non-cardiac Chest Pain (General disorders) | 4 (4)
Oral Dysesthesia (Gastrointestinal disorders) | 28 (43)
Oral Pain (Gastrointestinal disorders) | 11 (12)
Pain (General disorders) | 32 (58)
Palmer Plantar Erythrodysesthesia (Skin and subcutaneous tissue disorders) | 33 (82)
Rash (Skin and subcutaneous tissue disorders) | 33 (82)
Paresthesia (Nervous system disorders) | 17 (22)
Neuropathy (Nervous system disorders) | 4 (7)
Platelet Count Decrease (Investigations) | 23 (29)
Proteinuria (Renal and urinary disorders) | 39 (79)
Amylase Increase (Investigations) | 3 (3)
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 6 (7)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 11 (13)
Stomach Pain (Gastrointestinal disorders) | 3 (7)
Thromboembolic Event (Vascular disorders) | 3 (4)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 14 (21)
Weight Loss (Investigations) | 8 (12)
White Blood Cell Decrease (Investigations) | 29 (61)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-11): https://cdn.clinicaltrials.gov/large-docs/90/NCT01630590/Prot_SAP_000.pdf